CLINICAL TRIAL: NCT00235079
Title: Treatment and Prevention of Pericarditis With Colchicine. A Multicenter Double Blind Randomized Trial. The CORP 2 Trial: COlchicine for Recurrent Pericarditis.
Brief Title: Study of Colchicine to Treat and Prevent Recurrent Pericarditis After Failure of Conventional Treatment.
Acronym: CORP 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Sanitaria Locale 3, Torino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCASL30501-4; EUDRACT number 2005-001570-28
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Pericarditis; Recurrence
Keywords: Pericarditis; Recurrence; Therapeutics; Prevention; Colchicine
MeSH Terms: conditions — Pericarditis; Recurrence | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Experimental): Colchicine 0.5mg BID (>70Kg) or 0.5 once daily for 6 months
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo 0.5mg BID (>70Kg) or 0.5 once daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5mg BID (>70Kg) or 0.5 once daily for 6 months
  Arms: Colchicine
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether colchicine is safe and effective in treatment and prevention of recurrent pericarditis after failure of conventional treatment.

DETAILED DESCRIPTION:
Colchicine is safe and effective in the management of recurrent pericarditis after failure of conventional treatment. Preliminary data (observational, non-randomized studies without a control group) have shown that the drug may be effective in treatment of the second and subsequent recurrence and the prevention of further recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the second and subsequent attack of recurrent pericarditis,
* Age≥ 18 years,
* Informed consent.

Exclusion Criteria:

* Suspected neoplastic, tuberculous, or purulent etiology,
* Known severe liver disease and/or elevated transaminases >1.5 times the upper limit of normality,
* serum creatinine>2.5 mg/dl,
* Serum CK over the upper limit of normality or Known myopathy,
* Known gastrointestinal or blood disease,
* Pregnant or lactating women or women not protected by a contraception method,
* Known hypersensibility to colchicine,
* Treatment with colchicine at the enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at 18 months | 18 m onths

SECONDARY OUTCOMES:
Symptom persistence at 72 hours, remission rate at 1 week. Disease-related re-hospitalization, cardiac tamponade, constrictive pericarditis within the duration of the study. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Imazio, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital. ASL 3 Torino (Coordinating Center); Rita Trinchero, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital. ASL 3 Torino (Coordinating Center).
Locations (4):
- Italy (4):
  - Cardiology Department. Maria Vittoria Hospital ASL3 Torino (Coordinating Center), Torino, Torino
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Ospedale Regionale, Bolzano
  - Ospedale di Rivoli, Rivoli

REFERENCES:
- [Background] Imazio M, Cecchi E, Ierna S, Trinchero R; CORP Investigators. CORP (COlchicine for Recurrent Pericarditis) and CORP-2 trials--two randomized placebo-controlled trials evaluating the clinical benefits of colchicine as adjunct to conventional therapy in the treatment and prevention of recurrent pericarditis: study design and rationale. J Cardiovasc Med (Hagerstown). 2007 Oct;8(10):830-4. doi: 10.2459/JCM.0b013e3280110616. PMID 17885522
- [Derived] Imazio M, Belli R, Brucato A, Cemin R, Ferrua S, Beqaraj F, Demarie D, Ferro S, Forno D, Maestroni S, Cumetti D, Varbella F, Trinchero R, Spodick DH, Adler Y. Efficacy and safety of colchicine for treatment of multiple recurrences of pericarditis (CORP-2): a multicentre, double-blind, placebo-controlled, randomised trial. Lancet. 2014 Jun 28;383(9936):2232-7. doi: 10.1016/S0140-6736(13)62709-9. Epub 2014 Mar 30. PMID 24694983